CLINICAL TRIAL: NCT05190588
Title: Efficacy of Mesotherapy on Pain and Function in Patients With Knee Osteoarthritis
Brief Title: Efficacy of Mesotherapy in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Hakan Alkan, Clinical Professor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-60116787-020-63769
Record Dates: First submitted 2021-11-26; First posted 2022-01-13 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Mesotherapy

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled clinical study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (No Intervention): Quadriceps Strength 10 repetition in three-set, 5 times a week
- Mesotherapy (Active Comparator): Group 2: Mesotherapy (MT) Sterile and disposable (0.26mm × 4mm and 0.3mm × 13 mm, Terumo) will be used. Patients will receive 2 ml of 2% lidocaine, 2 ml of pentoxifylline and will be used. Injection techniques (IDP=2-4 MM) AND (IDS=1-2 MM) will be used. One time a week for a total of 3 times.
  Interventions: Other: Mesotherapy

INTERVENTIONS:
Other: Mesotherapy — Mesotherapy (MT) Sterile and disposable (0.26mm × 4mm and 0.3mm × 13 mm, Terumo) will be used. Patients will receive 2 ml of 2% lidocaine, 2 ml of pentoxifylline and will be used. Injection techniques (IDP=2-4 MM) AND (IDS=1-2 MM) will be used.
  Arms: Mesotherapy

SUMMARY:
Purpose: The investigators aimed to determine whether this treatment is effective on pain and function by applying mesotherapy treatment to patients followed up with gonarthrosis.

Methods: This study is a prospective randomized controlled study. The research will be carried out between November 2021 and April 2022 in Pamukkale University Physical Medicine and Rehabilitation (PMR) After the approval of the Pamukkale University Faculty of Medicine Ethics Committee, 38 patients diagnosed with gonarthrosis will be divided into 2 groups using a table of random numbers. The first group will be the group that only applied quadriceps strength exercise and Mesotherapy will be applied to the second group along with quadriceps strength exercise.

The data will be analyzed with the SPSS package program. Continuous variables will be given as mean ± standard deviation and categorical variables as numbers and percentages. parametric test Test of Significance of Difference Between Two Means in comparison of independent group differences when assumptions are met; When parametric test assumptions are not met, the Mann-Whitney U test will be used to compare independent group differences. In addition, the relationships between continuous variables will be examined with Spearman or Pearson correlation analyzes and the differences between categorical variables will be examined with Chi-square analysis. Since there is no similar study conducted and there is no possibility to conduct a pilot study, assuming that a moderate effect size will be obtained as a result of the power analysis made in the direction of the hypothetical expectations, it was taken to obtain 80% power with 95% confidence, and it was calculated that at least 38 people should be included in the study.

DETAILED DESCRIPTION:
Detailed Description:

This study is a prospective randomized controlled study. The research will be carried out in Pamukkale University Physical Medicine and Rehabilitation (PMR) After the approval of the Pamukkale University Faculty of Medicine Ethics Committee,38 participants will be admitted to Pamukkale University PMR clinic will be included in this study. Patients will be informed about the content, purpose, and application of the study and their written consent will be obtained.

Treatment Protocol 38 patients diagnosed with gonarthrosis will be divided into 2 groups using random numbers table. The first group will be the group that only applied quadriceps strength exercise and Mesotherapy will be applied to the second group along with quadriceps strength exercise.

Group 1: Exercise Group (Quadriceps Strength)10 repetition in three-set, 5 times a week for three weeks Group 2: Mesotherapy (MT) once a week for three weeks. Patients will receive 2 ml of 2% lidocaine, 2 ml of pentoxifylline will be used. Sterile and disposable (0.26mm × 4mm and 0.3mm × 13 mm, Terumo) will be used for mesotherapy. and injection techniques (IDP=2-4 MM) AND (IDS=1-2 MM) will be used.

Statistics The data will be analyzed with the SPSS package program. Continuous variables will be given as mean ± standard deviation and categorical variables as numbers and percentages. parametric test

Test of Significance of Difference Between Two Means in comparison of independent group differences when assumptions are met; When parametric test assumptions are not met, the Mann-Whitney U test will be used to compare independent group differences. In addition, the relationships between continuous variables will be examined with Spearman or Pearson correlation analyzes and the differences between categorical variables will be examined with Chi-square analysis. Since there is no similar study conducted and there is no possibility to conduct a pilot study, assuming that a moderate effect size will be obtained as a result of the power analysis made in the direction of the hypothetical expectations, it was taken to obtain 80% power with 95% confidence, and it was calculated that at least 38 people should be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as Knee Osteoarthritis according to ACR criteria

Exclusion Criteria:

* Smaller than 40 years old
* Those who give false and contradictory information,
* Those who are poorly oriented with cooperation, -Patients using non-steroidal anti-inflammatory, patients with a history of knee surgery, --
* Patients with meniscus lesions

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
VAS | 3 weeks
  Visual analogue scale (Total scale score can be ranged between 0 to 10. 0: no pain, 10:worst pain)

SECONDARY OUTCOMES:
WOMAC scale | 3 weeks
  Western Ontario and McMaster Universities Osteoarthritis Index (Test Questions are scored on a scale of 0-4 which correpond to: none(0), mild(1), moderate (2), severe (3) extreme (4). The scores for each subscales are summed up with a possible score 0-20 for pain, 0-8 for stiffness, 0-68 for physical function.)

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Sarsan, Principal Investigator — Pamukkale U
Locations (1):
- Pamukkale University, Denizli, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Felson DT, McLaughlin S, Goggins J, LaValley MP, Gale ME, Totterman S, Li W, Hill C, Gale D. Bone marrow edema and its relation to progression of knee osteoarthritis. Ann Intern Med. 2003 Sep 2;139(5 Pt 1):330-6. doi: 10.7326/0003-4819-139-5_part_1-200309020-00008. PMID 12965941
- [Background] Pelletier JP, Martel-Pelletier J, Abramson SB. Osteoarthritis, an inflammatory disease: potential implication for the selection of new therapeutic targets. Arthritis Rheum. 2001 Jun;44(6):1237-47. doi: 10.1002/1529-0131(200106)44:63.0.CO;2-F. No abstract available. PMID 11407681
- [Background] Felson DT, Chaisson CE, Hill CL, Totterman SM, Gale ME, Skinner KM, Kazis L, Gale DR. The association of bone marrow lesions with pain in knee osteoarthritis. Ann Intern Med. 2001 Apr 3;134(7):541-9. doi: 10.7326/0003-4819-134-7-200104030-00007. PMID 11281736
- [Background] Huang L, Guo B, Xu F, Zhao J. Effects of quadriceps functional exercise with isometric contraction in the treatment of knee osteoarthritis. Int J Rheum Dis. 2018 May;21(5):952-959. doi: 10.1111/1756-185X.13082. Epub 2017 May 25. PMID 28544687
- [Background] Kocak AO. Intradermal mesotherapy versus systemic therapy in the treatment of musculoskeletal pain: A prospective randomized study. Am J Emerg Med. 2019 Nov;37(11):2061-2065. doi: 10.1016/j.ajem.2019.02.042. Epub 2019 Feb 28. PMID 30876777